CLINICAL TRIAL: NCT01485016
Title: Observational Study Collecting Physiological and Biomechanical Data in Ambulatory Subjects With Epilepsy
Brief Title: Physiological and Biomechanical Data Collection Study in Epilepsy Subjects
Status: Completed | Type: Observational
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E-32
Record Dates: First submitted 2011-11-21; First posted 2011-12-05 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Epilepsy
Keywords: epilepsy; ECG; accelerometer
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ambulatory epilepsy subjects

SUMMARY:
The purpose of this study is to gather changes in physiological and biomechanical data during daily activity and sleep in epilepsy subjects.

DETAILED DESCRIPTION:
The purpose of this study is to gather changes in physiological and biomechanical data such as ECG, respiration, and accelerometry data during daily activity and sleep in pediatric and adult subjects with epilepsy. Subjects will use a device that enables monitoring of the human state in everyday, free-living environments.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be six (6) years of age or older
2. Subject has a clinical diagnosis of epilepsy
3. Subject is currently taking at least one antiepileptic medication.
4. Subject must be in good general health and fully ambulatory.
5. Subject or guardian must be willing and able to complete informed consent and/or assent for children and HIPAA authorization.

Exclusion Criteria:

1. Subjects with chest circumference smaller than 29 inches or greater than 47 inches.
2. Subjects with existing signs of skin irritation, rash, damage or infection on the torso that in the opinion of the investigator would prevent the subject's participation in the study.
3. Subjects with a medical condition that in the opinion of the investigator would affect his/her ability to participate in the study.
4. Subjects with implanted defibrillators, pacemakers or neurostimulators (e.g., vagus nerve stimulators or pain stimulators).
5. Subjects who are pregnant or lactating.
6. Subjects with severe psychiatric disease that in the opinion of the investigator would prevent the subject's successful completion of the study.
7. Subjects 6 to 16 years of age with moderate/severe learning difficulties or those who may be at risk of self-harm.
8. Subjects prescribed drugs specifically for a cardiac or autonomic disorder that in the investigator's opinion would affect heart rate response unless the patient has ictal tachycardia while taking said drugs. These include, but are not limited to, beta adrenergic antagonists ("beta blockers").
9. Subjects with cardiovascular arrhythmias or cardiac disease that would preclude the ability to detect intrinsic changes in heart rate due to activity, stress, or seizure. This would include but not be limited to chronic atrial fibrillation or chronotropic incompetence.
10. Subjects with a history of dependence on alcohol or narcotic drugs within the past 2 years as defined by DSM IV-R.
11. Subjects currently participating in another clinical study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric epilepsy patients willing to provide physiological and biomechanical data
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To gather changes in physiological and biomechanical data in epilepsy subjects | 72 hours
  The E-32 study was designed to capture the subject's physiological and biomechanical data such as ECG data and rate, respiratory data and rate, and body orientation, motion and movement (accelerometry) during typical events such as walking, sitting, running and sleeping in order to help build a database of stereotypical human activity.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Denham, DO, Principal Investigator — Clinical Trials of Texas, Inc.; Bryan Olin, Ph.D, Study Director — Cyberonics, Inc.
Locations (1):
- Clinical Trials of Texas, Inc., San Antonio, Texas, United States